CLINICAL TRIAL: NCT06210724
Title: Use of Faecal Biomarkers After Acute Diverticulitis: Can They Risk Stratify for Colorectal Cancer?
Brief Title: FIT in Diverticulitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Surrey County Hospital NHS Foundation Trust (Other)
Collaborators: GUTS - Fighting Bowel Cancer (Unknown); Minimal Access Therapy Training Unit (Other)
Responsible Party: Sponsor
Other Study IDs: 55623; 323724 (Other: IRAS); 55623 (Other: CPMS)
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-01

CONDITIONS: Diverticulitis; Colorectal Cancer
Keywords: Faecal Immunochemical test for haemoglobin; FIT; Faecal calprotectin; Faecal microbiome
MeSH Terms: conditions — Diverticulitis; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study cohort: In addition to standard of care, three faecal samples will be obtained. On as soon as possible after diagnosis, one at three weeks post diagnosis and one at six.
  Interventions: Diagnostic Test: Faecal immunochemical test for haemoglobin, faecal calprotectin, faecal microbiome

INTERVENTIONS:
Diagnostic Test: Faecal immunochemical test for haemoglobin, faecal calprotectin, faecal microbiome — Faecal samples to be collected by patients at home and delivered via post to a bowel cancer screening hub for analysis

SUMMARY:
Background and study aims

Diverticular disease or diverticulosis is a benign disease of the colon. Diverticulae are pockets of bowel wall which protrude through weaknesses in the muscular wall of the colon. The mechanisms leading to their formation remains unclear and is likely a complex interaction of multiple factors. For the majority of people these pockets are incidental findings they can become inflamed which is called diverticulitis.

The main aim of this study is to see if a faecal samples, which will be tested for hidden blood content with a faecal immunochemical test for haemoglobin (FIT), could be used as an alternative to currently used follow-up investigations for patients who have an episode of acute diverticulitis confirmed on a computerised tomography (CT) scan. These are colonoscopy, sigmoidoscopy or a special CT called CT colonoscopy.

The investigators will also be testing faecal calprotectin which is a marker of bowel inflammation and an assessment of the microbes that live in the bowel to see if this will provide further insights into the diagnosis and treatment of diverticulitis.

Who can participate?

All patients 18 or over admitted to a participating hospital with acute diverticulitis confirmed on a CT scan and who planned to have one of the currently used follow-up investigations are eligible.

What does the study involve?

The study will involve participants taking three stool (faecal) samples using faecal testing kits posted to participants. One is as close to their first solid stool after diagnosis as possible, the others are at 3 weeks after diagnosis and then 6 weeks after diagnosis.

What are the possible benefits and risks of participating?

There are no risks of participating. The investigators hope to demonstrate that a negative FIT test for patients after acute diverticulitis will be able to exclude a bowel cancer and prevent the majority of future patients having invasive and time consuming tests. There no additional benefit for participants for their current episode, as they will still need to have these tests.

Where is the study run from?

Royal Surrey County Hospital

When is the study starting and how long is it expected to run for?

09/10/2023-30/09/2024

Who is funding the study?

The study is being funded by MATTU (Minimal Access Therapy Training Unit), GUTS (GUTS - Fighting Bowel Cancer) and NHIR (National Institute for Health and Care Research).

Who is the main contact?

James Norman, On the study email rsch.colorectalDfitstudy@nhs.net

DETAILED DESCRIPTION:
What is the purpose of the study?

The main aim of this study is to see if a faecal immunochemical test (FIT), could be used as an alternative to currently used follow-up investigations, of colonoscopy, flexible sigmoidoscopy or CT (computerised tomography) colonography, for patients who have an episode of acute diverticulitis to exclude a colorectal cancer (CRC). As stated in the ASCPGBI consensus guidelines 2021 the risk of CRC in those with CT diagnosed uncomplicated diverticulitis is 1.6-1.9% and in those with complicated diverticulitis 7.8-10.9%.

Our primary aim is to determine whether single, or multiple faecal haemoglobin and faecal calprotectin results after an episode of acute diverticulitis can be used to risk stratify for further investigations to exclude colorectal cancer.

Our secondary aims are:

To determine whether single, or multiple faecal haemoglobin and faecal calprotectin results after an episode of acute diverticulitis could be used to risk stratify for further investigations to exclude other colonic findings such as high-risk adenoma?

Would including demographic factors such as age or anaemia allow better risk stratification?

Assess the faecal microbiome in patients with acute diverticulitis and how it changes as inflammation settles.

Any antibiotic treatment will also be recorded and the effect on the faecal microbiome analysed.

Inclusion criteria:

Computerised tomography diagnosis of acute diverticulitis Participants capable of giving informed consent Aged ≥ 18 years Planned for colonoscopy, flexible sigmoidoscopy or CT colonoscopy after diverticulitis diagnosis

Exclusion criteria:

Paediatric patients (<18 years) Not provided at least 1 FIT sample Unable to/unwilling to provide informed consent Withdrawal of consent for inclusion in study Previous pan-proctocolectomy, subtotal colectomy surgery, or presence of stoma Diagnosed with colorectal cancer Mental health illness limiting compliance Treated in hospital with colonic resection Did not have colonoscopy, flexible sigmoidoscopy or CT colonoscopy

Recruitment:

Patients who attend hospital with a diagnosis of acute diverticulitis confirmed on a CT scan and who have had a clinical decision to follow-up with either a colonoscopy, flexible sigmoidoscopy or CT colonography will be approached for written consent to participate.

Patients will then be posted a patient information leaflet and a pack with collection devices to take samples at home and post back. The results of their follow-up investigation (colonoscopy, flexible sigmoidoscopy or CT colonography + any histology) will be collected when completed

Involvement for patients will involve collecting and posting back in pre-paid envelopes faecal samples on their first solid stool (or as soon as possible after diagnosis) and at 3 and 6 weeks post-diagnosis.

Sample size: 275 - Estimated using available data on diverticulitis and stratified data from FIT use in 2WW patients.

ELIGIBILITY:
Inclusion Criteria:

* Computerised tomography diagnosis of acute diverticulitis
* Participants capable of giving informed consent
* Aged ≥ 18 years
* Clinical decision for colonoscopy, flexible sigmoidoscopy or CT colonoscopy follow-up after diverticulitis diagnosis

Exclusion Criteria:

* Paediatric patients (<18 years)
* Not provided at least 1 faecal sample
* Unable to/unwilling to provide informed consent
* Withdrawal of consent for inclusion in study
* Previous pan-proctocolectomy, subtotal colectomy surgery, or presence of stoma
* Currently being treated for colorectal cancer
* Mental health illness limiting compliance
* Treated in hospital with colonic resection
* Did not have colonoscopy, flexible sigmoidoscopy or CT colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending hospital with a radiological diagnosis of acute diverticulitis
Sampling Method: Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-28 (Estimated)

PRIMARY OUTCOMES:
Colorectal Cancer | Dependant on timing of investigation but expected 6-12 weeks
  Diagnosis or absence of colorectal cancer on follow-up investigation (Colonoscopy, flexible sigmoidoscopy or CT colonography)and subsequent histology results if applicable.

SECONDARY OUTCOMES:
High risk adenoma | Dependant on timing of investigation but expected 6-12 weeks
  Diagnosis or absence of high risk adenoma on follow-up investigation (Colonoscopy, flexible sigmoidoscopy or CT colonography)and subsequent histology results if applicable.
Diverticulitis | Dependant on timing of investigation but expected 6-12 weeks
  Diagnosis or absence of ongoing diverticular inflammation on follow-up investigation (Colonoscopy, flexible sigmoidoscopy or CT colonography)and subsequent histology results if applicable.
Perianal disease | Dependant on timing of investigation but expected 6-12 weeks
  Diagnosis or absence of perianal disease on follow-up investigation (Colonoscopy, flexible sigmoidoscopy or CT colonography)and subsequent histology results if applicable.
Inflammatory bowel disease | Dependant on timing of investigation but expected 6-12 weeks
  Diagnosis or absence of inflammatory bowel disease on follow-up investigation (Colonoscopy, flexible sigmoidoscopy or CT colonography)and subsequent histology results if applicable.
Microscopic colitis | Dependant on timing of investigation but expected 6-12 weeks
  Diagnosis or absence of microscopic colitis on follow-up investigation (Colonoscopy, flexible sigmoidoscopy or CT colonography)and subsequent histology results if applicable.

OTHER OUTCOMES:
FIT (Faecal Immunochemical Test for haemoglobin) test result | 6 weeks
  Results of the three FIT tests taken by the participant, ≥ 10 defined as FIT positive
Faecal calprotectin test result | 6 weeks
  Results of the three faecal calprotectin tests taken by the participant, ≥ 50 defined as positive
Faecal microbiome | 6 weeks
  Results of the microbiome run on the three faecal samples taken by the participant
Blood tests | Will happen before CT diagnosing diverticulitis
  Haemoglobin and mean cell volume from routine blood tests when patient attended

CONTACTS AND LOCATIONS:
Overall Officials: Sally Benton, FRCPath, Study Director — Royal Surrey NHS foundation trust; James Norman, BMBS, MRCP, Principal Investigator — Royal Surrey NHS foundation trust
Locations (1):
- Royal Surrey County Hospital, Guildford, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data will be anonymised before analysis and before any data is shared with other researchers